CLINICAL TRIAL: NCT00370578
Title: Aspiration Device Myocardial Infarction Trial
Brief Title: Aspiration Device in Myocardial Infarction Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaE064990ctil; Yoav Turgeman MD
Record Dates: First submitted 2006-08-09; First posted 2006-08-31 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2006-08

CONDITIONS: Angioplasty
Keywords: STEMI, THROMBUS, ASPIRATION DEVICE, NO REFLOW
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: repeated thrombus aspiration during primary PCI

SUMMARY:
Early promising data are published focusing on the role of manual thrombus aspiration devices in patients with ST segment elevation (STEMI).

The aim of our single center randomized study is to evaluate the early and late effect of thrombus aspiration device (AD) after every stage during Primary PCI in the set-up of STEMI population.

Our hypothysis is that preforming thrombus aspiration after every stage of primary PCI may give early and late advantages compared to the standard primary PCI technique.

DETAILED DESCRIPTION:
ADMIT-Randomized Single Center Study with two arms:

Standard PCI versus Primary PCI, using thrombus aspiration device after ever step of the procedure.

Issues to be examined are:

1. Immediate angiographic differences between the study arms. By evaluation of: TIMI FLOW GRADE,TIMI FRAME COUNT,MYOCARDIAL BLUSH GRADE. No reflow phenomenae,
2. Infarc size evaluated by serum markers and non invasive parameters
3. In hospital major adverse cardiac events
4. Major adverse cardiac events during 30& 180 days of follow up

ELIGIBILITY:
Inclusion Criteria:

* patients with STEMI<12 from synptoms onset
* eligble for primary PCI regardless of initial TIMI flow grade.
* patients for rescue PCI after failed thrombolysis will also be included

Exclusion Criteria:

* womwn with known pregnancy or who are lactating
* pts with allergy to aspirin, clopidogrel or heparin
* inability to obtain informed consent
* known existence of life threatening diseases with a life expectency less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Limitation of infarct size
Early and follow up related (MACE)-major adverse cardiac events

SECONDARY OUTCOMES:
Efficacy of using aspiration device after every stage of Primary angiplasty

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Turgeman, MD, Principal Investigator — Technion-school of medicine, Haifa, Israel
Locations (1):
- HaEmek Medical Center, Afula, Israel